CLINICAL TRIAL: NCT05406037
Title: Diagnostic Marker of Mucormycosis : Development and Evaluation of a Diagnostic Assay on a Cohort of Sera
Brief Title: Biomarkers for Invasive Mucormycosis
Acronym: BIM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Plateforme PAGés, Analyses Glycoconjugués (Unknown); Région Hauts de France, France (Unknown); SATT Nord (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021_0462; 2021-A03202-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-05-20; First posted 2022-06-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-01

CONDITIONS: Mucorales Infection; Mucormycosis
Keywords: Mucormycosis; Invasive fungal infection; Cell wall oligo/polysaccharides; Biomarkers
MeSH Terms: conditions — Mucormycosis; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with MM: Age : from 3 to 75 years old ;
  - Specific medical conditions : patient hospitalized in one of the departments of the University Hospital of Lille or Amiens, in whom the diagnosis of mucormycosis will have been made on the criteria below, with compatible clinical and radiological evolution :
  * conventional mycology data and/or
  * positive q-PCR and/or
  * pathology data confirmed by PCR;
  Interventions: Biological: Venous sample
- High-risk patients without MM (control group 1): Age : from 18 to 75 ;
  - Specific medical conditions : patients hospitalized at the University Hospital of Lille or Amiens for whom a diagnosis of candidiasis or invasive aspergillosis has been made according to specific classifications (EORTC/MSG criteria, AspICU criteria)
  Interventions: Biological: Venous sample
- Patients with another IFI (control group 2): * Age : from 18 to 75 ;
  * Specific medical conditions : patients undergoing assessment for haematopoietic stem cell transplantation, considered at risk of invasive fungal infection but for whom the pre-transplant assessment will have excluded an ongoing infection.
  Interventions: Biological: Venous sample

INTERVENTIONS:
Biological: Venous sample — at Day 0, Day 3, Day 7, Day 14, Day 28 (7 ml blood sample collecting on dry tube) D0 = Diagnostic day

SUMMARY:
Mucormycosis (MM) is one of the main invasive fungal infection (IFI), and is determined by filamentous fungi belonging to the order of Mucorales, with a mortality rate ranging from 20 to 60% according to localization. Prompt initiation of adequate antifungal therapy is critical for treating mucormycosis. Early diagnostic is therefore essential. The presence in the Mucorales' cell wall of uncommon monosaccharides open interesting perspectives for the development of specific diagnostic biomarkers.

This study evaluate a diagnostic test for mucormycosis in a cohort of patients with MM and in control groups (high-risk patients without MM and patients with another IFI).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age : Children and adults from 3 to 64 years old (18 to 64 for controls)
* In patients whose consent has been collected after information. In the case of children, information on the study will be given to the holders of parental authority and then to the child to obtain their consent.
* Patient social insured
* Specific medical conditions :

  1. For the case group :

     Any patient hospitalized in one of the departments of the University Hospital of Lille, in which the diagnosis of mucormycosis was conducted on the following criteria:
     * Conventional mycology data and / or
     * Positivity of q-PRC and / or
     * Anatomopathologic diagnosis Associated with a compatible clinical situation
  2. For the control group 1 Patient assessed for hematopoietic stem cell transplantation, considered at risk for IFI but for whom the pre-transplantation review will have excluded an ongoing infection
  3. For control group 2 Any patient hospitalized in a department of Lille University Hospital, in which the diagnosis of disseminated candidiasis or invasive pulmonary aspergillosis has been made according to specific classifications (EORTC/MSG criteria, AspICU criteria)

Exclusion Criteria:

* Patients for whom the inclusion criteria are not met
* Co-infection mucormycosis/other IFI

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients cared for at the University Hospitals of Lille and Amiens (France)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Values of the biomarker studied in the patient group versus control groups, expressed as Optical density (OD). | at Day 0
  Detection and quantification of the oligosaccharide biomarker will be performed using a sandwich type enzyme-linked immunosorbent assay (ELISA).Biomarker values could also be reported in arbitrary units / mL (plotting the calibration curve).

SECONDARY OUTCOMES:
Kinetics of the biomarker value measured for hospitalized patients, expressed as Optical density (OD). | at Day 3, Day 7, Day 14 and Day 28
  At each day of interest (at Day 3, Day 7, Day 14 and Day 28), values of OD obtained with an in-house immunoenzymatic sandwich microplate assay for the detection of a specific carbohydrate epitope of Mucorales will be reported for each sera.
Number of participant with unfavorable clinical evolution (death at D28) | at day 28
  Description of the clinical evolution (death or survival at D28) in parallel with the kinetic of the biomarker value

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie CORNU, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital of Lille, Lille, Hauts-de-France, France